CLINICAL TRIAL: NCT01291615
Title: Phase I Study of Gemcitabine or S-1 Adjuvant Therapy After Hemihepatectomy for Biliary Tract Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kansai Hepatobiliary Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHBO1003; UMIN000004682 (Registry Identifier: UMIN)
Record Dates: First submitted 2011-01-03; First posted 2011-02-08 (Estimated); Last update posted 2014-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; S 1 (combination); titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Gemcitabine group (Experimental): 800mg/m2 - 1000mg/m2, day 1 every 3 weeks. day 1, 15 every 4 weeks. day 1, 8 every 3 weeks. day 1, 8, 15, every 4 weeks
  Interventions: Drug: Gemcitabine
- S-1 group (Experimental): S-1 40mg/day - 120mg/day (depend on body surface area) day 1-14, every 3 weeks day 1-28, every 6 weeks
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: Gemcitabine — 800mg/m2 - 1000mg/m2, day 1 every 3 weeks. day 1, 15 every 4 weeks. day 1, 8 every 3 weeks. day 1, 8, 15, every 4 weeks
  Other Names: gemzer
  Arms: Gemcitabine group
Drug: S-1 — S-1 40mg/day - 120mg/day (depend on body surface area) day 1-14, every 3 weeks day 1-28, every 6 weeks.
  Other Names: TS-1
  Arms: S-1 group

SUMMARY:
To decide maximum tolerated dose and/or recommended dose of Gemcitabine or S-1 adjuvant therapy after hemihepatectomy

DETAILED DESCRIPTION:
There is no standard adjuvant therapy after liver hemi-hepatectomy due to bile duct cancer, because of high surgical morbidity ratio and high adverse event ratio of adjuvant therapy. For example, our preliminary results showed that regular gemcitabine administration (1000mg/m2, day1, 8, 15 every 4 weeks) after hemihepatectomy was too toxic and induced severe leukocytopenia and/or thrombocytopenia. Herein, we planned this study to decide more safety adjuvant protocol(recommend dose) for gemcitabine and S-1 after hemihepatectomy using continual reassessment method analysis. In this study, we decided that tolerable ratio of dose-limiting toxicity would be less than 10%.

ELIGIBILITY:
Inclusion Criteria:

1. Biliary tract cancer (>= UICC Stage IB)
2. R0 or R1 resection due to biliary tract cancer (BTC)
3. ECOG performance status must be 0 or 1
4. The patient underwent no other treatment than surgery for BTC
5. Neutrophil must be over 1500/μl, platelet must be over 100,000/μl, AST and ALT must be less than five times the normal limit, total bilirubin must be less than three times the normal limit, and creatinin must be less than 1.2 mg/dl.
6. The patient can intake drugs per os.
7. From 4 to 12 weeks after the surgery
8. Written informed consent

Exclusion Criteria:

1. Existence of active double cancer
2. The patient suffered from severe drug allergy
3. Sever complications (interstitial pneumonia, heart failure, renal failure, liver failure, ileus, incontrollable diabetes mellitus, and so on)
4. Any active infections exist.
5. Pregnancy
6. Severe mental disorder
7. Others

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-12; Primary Completion 2012-10 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
frequency in adverse events | up to 12 weeks
  The purpose of this study is to decide maximum tolerated dose and recommended dose. Recommended dose is a dose which would induce dose-limiting toxicity in 10% of participants. This will be calculated by continual reassessment method.

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Nagano, MD, PhD, Study Director — Osaka University Graduate School of Medicine
Locations (1):
- Osaka University, Graduate School of Medicine, Osaka, Japan

REFERENCES:
- [Background] Kobayashi S, Nagano H, Sakai D, Eguchi H, Hatano E, Kanai M, Seo S, Taura K, Fujiwara Y, Ajiki T, Takemura S, Kubo S, Yanagimoto H, Toyokawa H, Tsuji A, Terajima H, Morita S, Ioka T. Phase I study of adjuvant gemcitabine or S-1 in patients with biliary tract cancers undergoing major hepatectomy: KHBO1003 study. Cancer Chemother Pharmacol. 2014 Oct;74(4):699-709. doi: 10.1007/s00280-014-2543-4. Epub 2014 Jul 30. PMID 25074036